CLINICAL TRIAL: NCT04332328
Title: Study of Demographic and Dietary Profile in Patients With Ulcerative Colitis in Upper Egypt
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Snaa Mohammed Sayed Ali, SMSALI, Assiut University
Other Study IDs: 3032020
Record Dates: First submitted 2020-03-31; First posted 2020-04-02 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Diet in Ulcerative Colitis Patients
MeSH Terms: interventions — Diet

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ulcerative patients
  Interventions: Dietary Supplement: Diet
- Non ulcerative patients
  Interventions: Dietary Supplement: Diet

INTERVENTIONS:
Dietary Supplement: Diet — Group of diet types

SUMMARY:
Diet is known to play role in the complex etiology of UC.Patient with UC tend to adapt unguided dietary habits without the guidance of a dietician or physician (Dejong,M.J 2019).so identification of nutritional gaps is needed to facilitate the development of evidence-based dietary guideline and subsequently give correct dietary advice to UC patients(Haskkey,N et al 2017).

ELIGIBILITY:
Inclusion Criteria:

* patients with ulcerative colitis diagnosed by clinical Endoscopic and histopathological methods

Exclusion Criteria:

-

Patients with any co morbidity ( HTN,DM,Primary sclerosing cholangitis, as those patients need some restrictions of diet which may affect the prognosis of the disease)

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with ulcerative colitis with no other comorbidities
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2020-11-01 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Study of demographic and dietary profile in patients with ulcerative colitis in upper Egypt | A year
  Study of demographic and dietary profile in patients with ulcerative colitis in upper Egypt